CLINICAL TRIAL: NCT04960293
Title: "Comparison of Pain After Uterine Artery Embolization Using Spherical Gelfoam or Tris-acryl Gelatin Microsphere in Patients With Symptomatic Fibroids: A Prospective, Randomized Study
Brief Title: Spherical Gelfoam Versus Tri-acryl Microsphere for Uterine Artery Embolization for Symptomatic Fibroids
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4-2021-0467
Record Dates: First submitted 2021-06-23; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Symptomatic Uterine Fibroids
Keywords: Fibroid; Embolization; Pain; Inflammation
MeSH Terms: conditions — Leiomyoma; Pain; Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spherical gelfoam (Experimental): Patients who receive uterine artery embolization for symptomatic fibroids
  Interventions: Procedure: uterine artery embolization using spherical gelfoam
- Microsphere (Active Comparator): Patients who receive uterine artery embolization for symptomatic fibroids
  Interventions: Procedure: uterine artery embolization using tri-acryl gelatin microsphere

INTERVENTIONS:
Procedure: uterine artery embolization using spherical gelfoam — Uterine artery embolization is performed using spherical gelfoam. All other processes are same.
  Arms: Spherical gelfoam
Procedure: uterine artery embolization using tri-acryl gelatin microsphere — Uterine artery embolization is performed using tris-acryl gelatin microsphere. All other processes are same.
  Arms: Microsphere

SUMMARY:
The primary purpose of this study is to compare pain after uterine artery embolization using spherical gelfoam or tris-acryl gelatin microsphere in patients with symptomatic fibroids

DETAILED DESCRIPTION:
Uterine artery embolization(UAE) is a minimally invasive treatment alternative to hysterectomy and myomectomy in symptomatic fibroids. However, post-procedural pain after UAE remains a major problem. The spherical gelfoam and tri-acryl gelatin microsphere are two embolic materials used for UAE. Therefore, the aim of study is to compare pain intensity and inflammation after uterine artery embolization using the two embolic agents with symptomatic fibroids.

ELIGIBILITY:
Inclusion Criteria:

1. Women with symptomatic fibroids (age: 20 - 60 years old)

Exclusion Criteria:

1. Bradycardia (<45 bpm)
2. Conduction abnormalities
3. Liver failure
4. renal failure
5. Uncontrolled hypertension
6. High grade obesity (BMI ≥ 30 kg/m2)
7. Drug allergy
8. Illiteracy
9. Pregnancy

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Pain score (VAS score) | up to 24 hours after embolization
  Maximum pain score measured during 24 hours after embolization

SECONDARY OUTCOMES:
C-reactive protein (mg/L) | the day before and 24 hours after embolization
  inflammatory markers
Tumor necrosis rate after embolization | 1 day and 3 months after embolization
  technical success indicator
Symptom severity questionnaire | before and 3 months after embolization
  clinical success indicator
White blood cell count (/µL) | the day before and 24 hours after embolization
  inflammatory markers
Neutrophil percentage (%) | the day before and 24 hours after embolization
  inflammatory markers
Cumulative fentanyl dose (µg) | within 24 hours after embolization
  Total amount of IV fentanyl administered
Use of rescue analgesics (%) | within 24 hours after embolization
  Necessity of additional rescue analgesics
Lymphocyte percentage (%) | the day before and 24 hours after embolization
  Inflammatory marker

CONTACTS AND LOCATIONS:
Overall Officials: Man-Deuk Kim, Principal Investigator — Department of Radiology, Severance hospital
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided